CLINICAL TRIAL: NCT01367379
Title: The Effect of the Duty Loading on the Stress Response of Physician
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taipei City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 201104059RC
Record Dates: First submitted 2011-06-03; First posted 2011-06-07 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Physiological Stress; Psychological Stress
Keywords: Physician; duty loading; stress response; Physician with different amount of duty area
MeSH Terms: conditions — Stress, Psychological; Fractures, Stress | interventions — Blood Pressure Monitors; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Physician of internal medicine in Taipei city hospital
  Interventions: Procedure: 24 hour EKG and blood pressure monitor; Other: Blood and urine sampling

INTERVENTIONS:
Procedure: 24 hour EKG and blood pressure monitor — All subjects will have non-invasive 24 hour EKG and 24 hour EKG monitoring for 24 hours.
Other: Blood and urine sampling — Right before and after the duty loading, all subjects will have blood samplings, including CRP, WBC, IL-6, Fibrinogen, insulin, IL-6, Procalcitonin, TNF-alfa, catecholamine level. Right after the duty loading, all subjects will have urine samplings for cortisol and catecholamine level.(blood : 15CC/time and 2~4 times/month)

SUMMARY:
The investigators will study in the possibility of cardiovascular disease, caused by the duty loading, of physician of internal medicine. The investigators will also explore if there {dose response effect} between the duty loading and the stress response of physicians of internal medicine. Therefore, the investigators will compare the stress responses of physicians of internal medicine during with different duty loading ( non-duty day, one duty area with 3 wards, 2 duty areas with 6 wards) in a observational method. Those stress response will be measured by cardiovascular risk indicators, including blood pressure, heart rate variability, blood sampling and urine sampling.

ELIGIBILITY:
Inclusion Criteria:

* Attending physicians of internal medicine of Taipei municipal hospital, certified by Taiwan society of internal medicine.

Exclusion Criteria:

* thyroid dysfunction
* pregnancy, diabetes mellitus
* history of cardiovascular disease (stroke, coronary arterial disease, or myocardial infraction)
* current smokers, or
* taking sleeping pills or B-blocker

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Attending physicians of internal medicine of Taipei municipal hospital, certified by Taiwan society of internal medicine. We will compare those results of outcome variables of different amount of duty area.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The physiological change of physician during different duty loadings | 4 months
  The investigators will also explore if there {dose response effect} between the duty loading and the stress response of physicians of internal medicine, and will compare the stress responses of physicians of internal medicine during with different duty loading in a observational method. Those stress response will be measured by cardiovascular risk indicators, including blood pressure, heart rate variability, blood sampling and urine sampling.

CONTACTS AND LOCATIONS:
Overall Officials: Yue Leon Guo, Professor, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan university hospital, Taipei, Taiwan